CLINICAL TRIAL: NCT04118062
Title: Communicating With Patients on Cancer Resistance to Treatment: the Development of a Communication Tool. A Qualitative Cross-sectional Study of Professionals, Patients, Parents of Sick Children, and Expert Patients, in the Context of Triple Negative or Luminal B Breast Cancer, Metastatic Uveal Melanoma and Pediatric Cancers.
Brief Title: Communicating With Patients on Cancer Resistance to Treatment: the Development of a Communication Tool. (HECTOR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IC 2018-09
Record Dates: First submitted 2019-09-11; First posted 2019-10-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Uveal Melanoma; Triple Negative Breast Cancer; Luminal B Breast Cancer; Pediatric Cancer
MeSH Terms: conditions — Uveal Melanoma; Triple Negative Breast Neoplasms; Neoplasms | interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Intervention Model Description: To meet our objectives, the research team has developed a cross-sectional and mixed exploratory research according to three successive steps :
  Step 1: Questionnaires and semi-structured individual interviews will : (a) to identify patients' needs and (b) to build the initial contents of the tool, items and issues. Four patients' populations will be recruited in this step : metastatic uveal melanoma, triple negative breast cancer, luminal B breast cancer, and pediatric cancer. This step will be conducted in parallel with these populations.
  Step 2 : Focus groups : to evaluate the acceptability and applicability of the tool in this clinical context with expert patients, researchers and clinicians.
  Step 3 : The DELPHI consensus method : to validate the contents of the booklet for patients with expert patients, researchers and clinicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Metastatic Uveal Melanoma (Other): Questionnaires and semi-structured individual interviews with patients with Metastatic Uveal Melanoma
  Interventions: Behavioral: Questionnaires; Behavioral: Semi-structured individual interviews
- Triple Negative Breast Cancer (Other): Questionnaires and semi-structured individual interviews with patients with Triple Negative Breast Cancer
  Interventions: Behavioral: Questionnaires; Behavioral: Semi-structured individual interviews
- Luminal B Breast Cancer (Other): Questionnaires and semi-structured individual interviews with patients with Luminal B Breast Cancer
  Interventions: Behavioral: Questionnaires; Behavioral: Semi-structured individual interviews
- Pediatric Cancer (Other): Questionnaires and semi-structured individual interviews with parents of children with cancer.
  Interventions: Behavioral: Questionnaires; Behavioral: Semi-structured individual interviews
- Expert Patients (Other): Focus groups (or group interviews) and DELPHI consensus method with expert patients
  Interventions: Other: Focus Group; Other: DELPHI Consensus Method
- Researchers and Clinicians (Other): Focus groups (or group interviews) and DELPHI consensus method with Researchers and Clinicians
  Interventions: Other: Focus Group; Other: DELPHI Consensus Method

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires
  Arms: Luminal B Breast Cancer; Metastatic Uveal Melanoma; Pediatric Cancer; Triple Negative Breast Cancer
Behavioral: Semi-structured individual interviews — Semi-structured individual interviews
  Arms: Luminal B Breast Cancer; Metastatic Uveal Melanoma; Pediatric Cancer; Triple Negative Breast Cancer
Other: Focus Group — Focus Group
  Arms: Expert Patients; Researchers and Clinicians
Other: DELPHI Consensus Method — DELPHI Consensus Method
  Arms: Expert Patients; Researchers and Clinicians

SUMMARY:
Resistance to treatment is one of the major themes in cancer research. Despite this, the definition and clinical implications of resistance to treatment remain under-explored, and patient-physician communication in this context still constitutes a challenge. When resistance to cancer treatments occurs, physicians not only have to explain to the patient the phenomenon of resistance, often based on complex results (biological results, genomic tests, imaging, etc.), but also need to offer alternative therapies, whilst fostering shared medical decision-making. These different tasks are particularly challenging for clinicians, especially since there are large individual differences at patient level. Indeed, each patient has his or her own unique information needs, capacity for understanding, and level of desire to participate in treatment decisions.

DETAILED DESCRIPTION:
Although a challenge, better communicating around resistance to treatment carries many potential benefits. Indeed, in similar contexts of announcement of bad news and choice of care, Parker and collaborators (1) have highlighted the positive impact of individualized care, respecting the needs, quality of care, and quality of life of patients. Given the clinical stake, and the lack of scientific knowledge devoted to communication in the context of resistance to treatment, it appears necessary to better understand its modalities. In this perspective, research has proven the value of tools for supporting communication, including the issue of question booklets for patients. These tools provide patients with a list of questions submitted to them before the medical consultation, and which they can ask during the consultation, and throughout the treatment. This tool fosters communication by helping the patient obtain a level of information that is adapted to his or her needs and experience, and thus, to be better prepared for care. Despite significant interest for these booklets in the field of oncology, none has yet been developed in the specific context of resistance to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  1. To be 18 years of age or older ;
  2. To have metastatic uveal melanoma (MUM) or triple negative or luminal B breast cancer ;
  3. To have received the information that the disease is resistant to treatment ;
  4. To have read the information and signed the informed consent.
* Parents of a sick child:

  1. To be a parent (parental authority holder) of a child with cancer ;
  2. To have received the information that the child disease is resistant to treatment ;
  3. To have read the information and signed the informed consent.
* Expert patients:

  1. To be 18 years of age or older ;
  2. To have had cancer (regardless the cancer site) ;
  3. To participated to an expert patient training (fine knowledge of the illness, experience with the disease) ;
  4. To have read the information and signed the informed consent.
* Professionals:

  1. To be an oncologist (medical oncologist, surgeon, radiotherapist, supportive care specialist) and/or to be a researcher in oncology (doctor, biologist, geneticist ...) ;
  2. To have patients with a triple-negative or luminal B breast cancer or metastatic uveal melanoma which is resistant to anti-tumor treatments and/or to take part to a research on resistance to cancer treatment;
  3. To have read the information and signed the informed consent.

Exclusion Criteria:

* Patients & parents of a sick child:

  1. To have difficulties in understanding the French language.
  2. Have or have had cancer (criteria only for parents);
  3. Pregnant woman, likely to be pregnant or breastfeeding (criteria only for patients).
  4. Persons deprived of their liberty or under guardianship;
  5. Impossibility of study requirements respect for geographical, social or psychological reasons.
* Expert patients:

  1. To have difficulties in understanding the French language ;
  2. Currently being undergoing anti-tumor treatment.
* Professionals:

  1. To have difficulties in understanding the French language ;
  2. Not to be confronted in professional practice with resistance to anti-tumor treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2024-05-26 (Actual)

PRIMARY OUTCOMES:
List of patients' needs, particularly regarding communication with physicians | 18 months
  List of patients' needs in support, and information delivered by physicians in consultation
Items of communication booklet | 18 months
  Number and content of items, number of categories / themes,
Acceptability of the booklet evaluated | 18 months
  Items and issues revised and reformulated by the experts. Application of the booklet in the determined clinic: Modes of administration of the booklet and patients concerned identified. Implementation of the tool and relevant patients identified
Content of communication booklet validated | 18 months
  Consensus criteria: Consensus can be considered to have been reached if the majority of participants (70% or more) rank an item similarly

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie DOLBEAULT, PHD, Study Director — Institut Curie; Anne BREDART, PHD, Study Director — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets with interested reserachers, educators or clincians. Materials generated under the project will be disseminated in accordance with Institut Curie policies.
Time Frame: Data requests can be submitted starting 9 months after article publication and will made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Derived] Rault A, Dolbeault S, Terrasson J, Bouleuc C, Cottu P, Piperno-Neumann S, Rodrigues M, Vaflard P, Bredart A. Facilitating patient-oncologist communication in advanced treatment-resistant cancer: development and feasibility testing of a question prompt list. Pilot Feasibility Stud. 2024 Aug 28;10(1):116. doi: 10.1186/s40814-024-01543-y. PMID 39198868
- [Derived] Bredart A, Rault A, Terrasson J, Seigneur E, De Koning L, Hess E, Savignoni A, Cottu P, Pierga JY, Piperno-Neumann S, Rodrigues M, Bouleuc C, Dolbeault S. Helping Patients Communicate With Oncologists When Cancer Treatment Resistance Occurs to Develop, Test, and Implement a Patient Communication Aid: Sequential Collaborative Mixed Methods Study. JMIR Res Protoc. 2022 Jan 12;11(1):e26414. doi: 10.2196/26414. PMID 35019850